CLINICAL TRIAL: NCT02886871
Title: Mobile Phone-Based Physical Activity Intervention on University Staff
Brief Title: CalFitness Smartphone-Delivered Physical Activity Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Principal Investigator, Anil Aswani, Assistant Professor, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-03-8609-1
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Sedentary Lifestyle; Physical Activity
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Personalized Steps Goal (Experimental): Step Goal Delivery by Smartphone
  Interventions: Behavioral: Step Goal Delivery by Smartphone
- Constant Steps Goal (Active Comparator): Step Goal Delivery by Smartphone
  Interventions: Behavioral: Step Goal Delivery by Smartphone

INTERVENTIONS:
Behavioral: Step Goal Delivery by Smartphone

SUMMARY:
The overall goal of this study is to test personalized mobile phone-based physical activity interventions among staff members at the University of California, Berkeley. Most physical fitness applications for smartphones and activity trackers use a constant goal for the number of steps each day. However, if the step goals are dynamically adjusted according to past behavior, then the corresponding goals may encourage individuals to increase their physical activity level. This study consists of a randomized controlled trial in which we are assessing the efficacy of two different algorithms for calculating personalized goals for the number of steps each day.

ELIGIBILITY:
Inclusion Criteria:

* intent to become physically active
* own an iPhone
* willing to keep the iPhone in pockets during the day
* willing to install and use the intervention app every day for 4 months
* ability to speak and read English.

Exclusion Criteria:

* known medical conditions or physical problems that require special attention in an exercise program
* planning an international trip during the next 4 months, which could interfere with daily server uploads of mobile phone data
* pregnant/gave birth during the past 6 months
* severe hearing or speech problem
* history of an eating disorder
* current substance abuse
* current participation in lifestyle modification programs or research studies that may confound study results
* history of bariatric surgery or plans for bariatric surgery in the next 12 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Daily Steps Taken Per Day | 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Berkeley, Berkeley, California, United States

REFERENCES:
- [Derived] Zhou M, Fukuoka Y, Mintz Y, Goldberg K, Kaminsky P, Flowers E, Aswani A. Evaluating Machine Learning-Based Automated Personalized Daily Step Goals Delivered Through a Mobile Phone App: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2018 Jan 25;6(1):e28. doi: 10.2196/mhealth.9117. PMID 29371177